CLINICAL TRIAL: NCT04259333
Title: Celecoxib vs. Acetaminophen-codeine-caffeine for Postoperative Pain in Primary Elective Open Septorhinoplasty With Osteotomies: a Randomized Controlled Trial.
Brief Title: Celecoxib vs. Acetaminophen/Codeine/Caffeine for Post-operative Analgesia in Rhinoplasty.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blake Raggio (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Blake Raggio, Clinical Fellow, Humber River Hospital
Organization: Humber River Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16511
Record Dates: First submitted 2020-01-30; First posted 2020-02-06 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Pain, Postoperative; Surgery--Complications; Opioid Analgesic Adverse Reaction; Opioid Use
Keywords: opioid; rhinoplasty; pain, postoperative; celecoxib
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib; acetaminophen, codeine drug combination; Acetaminophen

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The surgeon (Care provider) performing all of the septorhinoplasty procedures will be blinded as to which pain medication the patients will receive postoperatively.
  The outcomes assessor evaluating the severity of bruising (using postoperative photographs taken on day of cast removal) will be blinded as to which pain medication the patient received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test Arm (Experimental): celecoxib 200 mg tablet by mouth every 12 hours for 7 days postoperatively prn pain
  Interventions: Drug: Celecoxib 200mg
- Control Arm (Active Comparator): codeine 30mg-acetaminophen 300mg-caffeine 15 mg tabelt by mouth every 4 hours for 7 days postoperatively prn pain
  Interventions: Drug: Acetaminophen, Codeine Drug Combination

INTERVENTIONS:
Drug: Celecoxib 200mg — Celecoxib tablet
  Other Names: celebrex
  Arms: Test Arm
Drug: Acetaminophen, Codeine Drug Combination — acetaminophen-codeine-caffeine tablet
  Other Names: tylenol #3
  Arms: Control Arm

SUMMARY:
The primary aim of this study is to evaluate whether celecoxib (CELEBREX) is equivalent to acetaminophen-codeine-caffeine (TYLENOL# 3) for the management of pain after primary elective open septorhinoplasty with osteotomies.

Secondary objectives include comparison of adverse medication effects and complications (e.g., bleeding events and bruising) that occur postoperatively.

Half of the study participants will receive celecoxib, and half will receive acetaminophen-codeine-caffeine.

We hypothesize that both interventions will exhibit no difference in pain control or postoperative bleeding, but that participants taking CELEBREX will experience less medication-related side effects and less bruising postoperatively.

DETAILED DESCRIPTION:
The recent recognition of the opioid crisis has prompted a nationwide search for alternative postoperative analgesia regimens, especially in the field of plastic and reconstructive surgery where patients exhibit a significant risk of persistent opioid use afterward.

As such, the contemporary facial plastics literature has noticed a surge in publications that implement various multi-modal analgesia (MMA) regimens to mitigate narcotic use postoperatively, the results of which seem promising.

Among the opioid-sparing medications utilized in MMA regimens, the selective COX-2 inhibitors (e.g., celecoxib, parecoxib) are of interest given their similar analgesic efficacy and decreased risk profile (less nausea, constipation, and dependence) compared to opioids. Furthermore, selective COX-2 inhibitors avoid adverse gastrointestinal and renal events, as well as the antiplatelet effects associated with conventional NSAIDs (e.g., ibuprofen and naproxen). For these reasons, selective COX-2 inhibitors make for the ideal analgesic to use after facial plastic surgery procedures, where increased bleeding can delay wound healing (e.g., increased bruising and swelling) and cause potentially devastating complications (e.g., hematoma after a facelift, or epistaxis after septorhinoplasty). Nonetheless, studies evaluating the role of selective COX-2 inhibitors as safe and effective alternatives to opioids in plastic surgery are scant.

The primary aim of this study is to evaluate whether celecoxib is equivalent to a routinely prescribed analgesia, acetaminophen-codeine-caffeine (trade name TYLENOL#3) for the management of pain after primary cosmetic open septorhinoplasty with osteotomies. Secondary objectives include comparison of adverse effects that occur post-operatively, with attention to medication side effects, as well as bleeding events and bruising.

We hypothesize that both interventions will exhibit no difference in pain control or postoperative bleeding or bruising, but that participants taking acetaminophen/codeine will experience more adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* • Patients 18-80 years old undergoing elective primary open septorhinoplasty with osteotomies by single surgeon, JA.

Exclusion Criteria:

* • Patients who undergo a rhinoplasty requiring a rib, ear, or temporalis fascia graft (confounding variables for the level of pain experienced)

  * Patients with a known history of chronic pain disorder, or who have gastrointestinal bleeds, peptic ulcer disease or who have other comorbidities that may prevent them from taking NSAIDs such as CELEBREX.
  * Patients with a history of radiation, active head and neck malignancy or other chronic pain disorders such as various rheumatologic diseases will be excluded to decrease confounding factors in assessing pain.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | until the time of cast removal (up to 8 days postoperatively)
  Difference in daily mean pain intensity based on Numeric Rating Scale (NRS). The NRS is composed of 0 (no pain at all) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Medication-related side effects | for side effects experienced up to the day of cast removal (up to 8 days postoperatively)
  patient self-reported questionnaire
Complications postoperatively | for complications experienced up to the day of cast removal (up to 8 days postoperatively)
  patient self-reported questionnaire
Bruising | day 6-8. depending on day of cast removal
  blinded outcome assessor will rank bruising severity based on Numeric Rating Scale (NRS), using postoperative photographs taken on day of cast removal. The NRS is composed of 0 (no brusing at all) to 10 (worst imaginable bruising).

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Asaria, MD, Principal Investigator — University of Toronto | FACE Cosmetic Surgery Toronto
Locations (1):
- FACE Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requests will be required to sign a Data Access Agreement

DOCUMENTS (1):
  • Informed Consent Form (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT04259333/ICF_000.pdf